CLINICAL TRIAL: NCT01861327
Title: The Use of Carbon Dioxide as a Contrast Media for Performing Endovascular Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nelson Wolosker (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor-Investigator, Nelson Wolosker, MD, PHD, Hospital Israelita Albert Einstein
Organization: Hospital Israelita Albert Einstein (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO2
Record Dates: First submitted 2013-02-26; First posted 2013-05-23 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Critical Lower Limb Ischemia; Abdominal Aortic Aneurysms
Keywords: Carbon dioxide; aortic aneurysm; angioplasty; Critical lower limb ischemia
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- lower limb angioplasty with CO2 (Experimental): lower limb angioplasty made with carbon dioxide as contrast media
  Interventions: Drug: CO2
- lower limb angioplasty with Iodine (Active Comparator): lower limb angioplasty made with Iodine as contrast media
  Interventions: Drug: Iodine contrast media
- aorto-iliac angioplasty with CO2 (Experimental): aorto-iliac angioplasty made with carbon dioxide as contrast media
  Interventions: Drug: CO2
- aorto-iliac angioplasty with Iodine (Active Comparator): aorto-iliac angioplasty made with Iodine as contrast media
  Interventions: Drug: Iodine contrast media
- endovascular AAA correction with CO2 (Experimental): endovascular abdominal aortic aneurysm (AAA) correction made with carbon dioxide as contrast media
  Interventions: Drug: CO2
- endovascular AAA correction with Iodine (Active Comparator): endovascular abdominal aortic aneurysm (AAA) correction made with Iodine as contrast media
  Interventions: Drug: Iodine contrast media

INTERVENTIONS:
Drug: CO2 — carbon dioxide (CO2) as arterial contrast media
  Arms: aorto-iliac angioplasty with CO2; endovascular AAA correction with CO2; lower limb angioplasty with CO2
Drug: Iodine contrast media — Iodine as arterial contrast media
  Arms: aorto-iliac angioplasty with Iodine; endovascular AAA correction with Iodine; lower limb angioplasty with Iodine

SUMMARY:
Prospective randomized comparison between endovascular procedures performed with iodinated contrast or carbon dioxide as intraarterial contrast.

DETAILED DESCRIPTION:
120 patients will undergo endovascular procedures: 40 for the treatment of lower limb ischemia caused by aortoiliac stenosis classified according to the consensus for the management of peripheral arterial disease (TASC) A or B with an indication for angioplasty as the inclusion criteria; 40 for the treatment of lower limb ischemia due to stenosis femoropopliteal TASC A or B with an indication of angioplasty as the inclusion criteria and 40 for the treatment of abdominal aortic aneurysm (AAA) with indication for endovascular repair. Of these procedures, half chosen randomly by computerized simple random, will be submitted to the endovascular procedure in question using only iodinated contrast and the other half will be submitted to the endovascular procedure using carbon dioxide (CO2). There will be no CO2 injection in the aortic arch or cerebral territory. The patient previously evaluated at the Hospital Municipal Dr. Moses Deutsch will be referred to the operating room of the Albert Einstein Hospital where it will be performed under general anesthesia with intubation or blockage associated with sedation, and the same in the supine position (DDH).The femoral artery will be punctured with Seldinger technique unilaterally or bilaterally, according to the indication for the procedure. By using the guide wire will be one or two sheaths inserted in a retrograde manner. Through the introducer, is manually injected retrogradely 50 ml of CO 2, in obtaining images of the apparatus module CO2 Philips mode subtraction angiography. In angioplasty for obstructive disease, with the module roadmap will be held the passage of the guidewire through the stenotic region or occlusion, and dilatation balloon angioplasty specific. After angioplasty, there will be a new injection of contrast for the evaluation of partial results. As appropriate, will be held stent placement, in which case there will be a last angiography with 50 ml of CO2. In endovascular repair of abdominal aortic aneurysms, there will be a first injection of CO2 for the study of the neck of the aneurysm and stent implantation. After the release of the entire stent, a new angiography is performed by injection of CO2 for the control of surgical outcome. In all procedures will be performed to measure pressure through the femoral sheath prior to angioplasty, after angioplasty and stent after the placement. During the use of CO2 as contrast medium, with questions at the trial of such factors as the extent of injury, indication of repair, endoleak, leak, rupture or thrombosis by arteriography will be performed by manual injection of iodinated contrast.Of course this amount of contrast is measured.

ELIGIBILITY:
Inclusion Criteria:

* critical lower limb ischemia resulting from arterial disease morphology TASC A or B or abdominal aortic aneurysms with correction indication
* Agreement and signing the informed consent.

Exclusion Criteria:

* exhibited severe chronic obstructive pulmonary disease (COPD)
* kidney failure
* heart failure
* pregnancy
* TASC C or D lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Contrastation analysis of the arterial lumen on endovascular procedures using CO2 as contrast media. | within 2 weeks of the procedure done we will analyze the quality of the images with CO2 and iodine contrast
  image evaluated ranging from 1 (poor -when there was significant loss of definition in the vessels and/or collateral circulation which precluded the procedure), 2 (fair - when there was some loss of definition in the vessels and/or collateral circulation but not impossible to perform the procedure) and 3 (good - when there was good contrast in the vessels and collateral circulation).

SECONDARY OUTCOMES:
clinical outcome: changes in the post-surgery ABI | within 24h of the procedure
  Identify changes in ankle-braquial index (ABI) after the procedures

OTHER OUTCOMES:
post surgery creatinin clearance measure by the Cockcroft and Gault equation | within 30 days of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil